CLINICAL TRIAL: NCT02103491
Title: Effects of Oral Salt Supplementation on Physical Performance During a Half-ironman
Acronym: SALTED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Camilo Jose Cela University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UCJC-14
Record Dates: First submitted 2014-03-26; First posted 2014-04-04 (Estimated); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Hyponatremia
Keywords: Half-ironman; Triathlon; Salt; Exercise; Performance
MeSH Terms: conditions — Hyponatremia; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Salt administration (Active Comparator): Participants were provided with 3 plastic bags each one containing 4 white capsules (e.g., a total of 12 capsules). In the salt group, the capsules were filled with a commercially available product that contains buffered electrolyte salts (Saltstick caps, Saltstick, California US). The total amount of electrolytes provided in the salt group was: 2580 mg of sodium (113 mmol), 3979 mg of chloride (112 mmol), 756 mg of potassium (19.3 mmol) and 132 mg of magnesium (5.4 mmol).
  Interventions: Dietary Supplement: Salt administration
- Placebo administration (Placebo Comparator): In the control group, participants received the same number of capsules with the exact same appearance but filled with an isocaloric placebo (cellulose).
  Interventions: Dietary Supplement: Placebo administration

INTERVENTIONS:
Dietary Supplement: Salt administration — Participants were provided with 3 plastic bags each one containing 4 white capsules (e.g., a total of 12 capsules). In the salt group, the capsules were filled with a commercially available product that contains buffered electrolyte salts (Saltstick caps, Saltstick, California US). The total amount of electrolytes provided in the salt group was: 2580 mg of sodium (113 mmol), 3979 mg of chloride (112 mmol), 756 mg of potassium (19.3 mmol) and 132 mg of magnesium (5.4 mmol). In the control group, participants received the same number of capsules with the exact same appearance but filled with an isocaloric placebo (cellulose). All the participants were instructed to ingest the contents of the first bag in the transition between the swimming and cycling sections, the second bag around the middle of the cycling leg and the third bag during the transition between the cycling and running sections.
  Arms: Salt administration
Dietary Supplement: Placebo administration
  Arms: Placebo administration

SUMMARY:
Background: Ultradistance athletes frequently consume salt supplements during competitions to compensate the loss of electrolytes by sweating. The aim of this study was to investigate the effectiveness of oral salt supplementation to improve exercise performance during a half-ironman triathlon. Methodology: Twenty-six experienced triathletes were matched for age, anthropometric data and training status and randomly placed into the salt group (113 mmol Na+ and 112 mmol Cl-) or the control group (cellulose). The experimental treatments were provided in unidentifiable capsules and were ingested before and during the race. Participants competed in a real half-ironman triathlon and race time was measured by means of chip timing. Pre and post-race, body mass, maximal force during a whole-body isometric strength test, maximal height during a countermovement jump, and blood samples were obtained. Sweat samples were obtained during the running section.

DETAILED DESCRIPTION:
Participants Forty healthy and well-trained triathletes were recruited by email or through internet announcements to participate in this study. Before enrolling in the investigation, a questionnaire about their medical history, previous training, previous triathlon experience and best race time in half-ironman triathlon races was filled out by each participant. Potential participants with a previous history of muscle disorder, cardiac or kidney disease or those taking medicines during the two prior weeks were discarded. Finally, twenty-six participants were selected and matched (in pairs) for age, anthropometric data, training and best race time. Then, an equal number of triathletes (n = 13) was randomly assigned to the control group or to the salt ingestion group. Main morphological variables, training status and best performance time in the half-ironman distance were similar between these groups (P > 0.05; Table 1). All the participants were informed of the risks and discomforts associated with the experiments and signed a written consent before their participation in this investigation. The study was approved by the Camilo Jose Cela Ethics Committee in accordance with the latest version of the Declaration of Helsinki.

Experimental Protocol Participants were instructed to perform light exercise and to avoid pain-relieving strategies (e.g., analgesic medications, manual massage, ice, etc) the two days before the race. In addition, participants were instructed to avoid any sources of caffeine and alcohol 24 h before the onset of the race. Three hours before the race, participants arrived at an area close to the start line having drunk 500 mL of tap water two hours before arrival. Participants had their habitual pre-competition meal and it was not standardized among participants to avoid affecting participants' pre-competition routines. However, the pre-competition meals were analyzed afterwards and their content in carbohydrates, proteins and salt was similar between groups.

On arrival, participants rested for 10 minutes in a recumbent chair and a 5-mL venous blood sample was drawn from an antecubital vein. The blood was allowed to clot and centrifuged at 5000g to obtain serum. Participants then completed a 10-min standardized warm-up consisting of running, dynamic leg exercises and practice jumps. After that, participants performed two countermovement vertical jumps (CMJ) for maximal height on a force platform (Quattrojump, Kistler, Switzerland) to assess pre-race leg power output. On command, the participant flexed their knees and jumped as high as possible while maintaining the hands on the waist and landed with both feet. The highest values for jump height and the peak muscle leg power during the concentric phase of the jump were used for statistical analysis. Participants were previously familiarized with the jump test.

After that, whole-body isometric muscle strength was measured by means of a hand-held pull gauge (Isocontrol Isométrico, EV-Pro, Spain) set at a frequency of 1000 Hz. For this measurement, participants stand on a 50 × 50 cm iron base connected to a handle-bar by a non-elastic cable. The isometric gauge was inserted within the cable and the height of the cable was individually set to provide a 135º knee flexion while the back and the arms were completely extended. Participants were instructed to perform a maximal pull by for 3-s using their whole body (mainly legs and arms) while maintaining this position. Verbal motivation was provided during the test. An adjustable lumbar-back protector was used for support and protection during the execution. Maximal and mean isometric strength were obtained during the test. Participants were previously familiarized with this measurement.

After that, participants were provided with 3 plastic bags each one containing 4 white capsules (e.g., a total of 12 capsules). In the salt group, the capsules were filled with a commercially available product that contains buffered electrolyte salts (Saltstick caps, Saltstick, California US). The total amount of electrolytes provided in the salt group was: 2580 mg of sodium (113 mmol), 3979 mg of chloride (112 mmol), 756 mg of potassium (19.3 mmol) and 132 mg of magnesium (5.4 mmol). In the control group, participants received the same number of capsules with the exact same appearance but filled with an isocaloric placebo (cellulose). All the participants were instructed to ingest the contents of the first bag in the transition between the swimming and cycling sections, the second bag around the middle of the cycling leg and the third bag during the transition between the cycling and running sections. This schedule was used to facilitate ingestion and electrolyte absorption during the race. Participants received a sample of these capsules (filled with placebo) the week before the race to practice the ingestion protocol during the transition and the cycling sector. Participants were encouraged to ingest all the capsules in the programmed schedule and to report any incidence during the capsule ingestion throughout the race.

Just 15-min before the race (and after their habitual warm-up), participants were weighed in their competition clothes (without wetsuit) and a segmental bioelectrical impedance analysis was performed (BC-418, Tanita, Japan) to predict pre-to-post race total body water changes. The race started at 12:00 h and consisted of 1.9 km of swimming, 75 km of cycling (1100 m net increase in altitude) and 21.1 km of running. Environment conditions were recorded at 30-min intervals and mean ± SD (range) dry temperature during the event was 22.5 ± 2.7ºC (18.8 - 26.6 ºC) with a relative humidity of 36.8 ± 8.3% (32 - 45%). The swim section was performed in a natural lake with water temperature at 17.5 ± 0.3ºC. All participants wore a neoprene wetsuit during the swim section. Participants drank and consumed food ad libitum and swam, cycled and ran at their own pace with no instructions given by the experimenters (apart from those related to capsule ingestion).

During the second transition (between the cycling and running legs), two sweat patches (Tegaderm+Pad, 3M, US) were placed on the forearm to collect sweat samples. For this purpose, participants went to an area located just outside the transition area and the forearm skin was cleaned with distilled water and alcohol and dried with clean gauze to eliminate any remains of previous sweat from the skin. After this, the sweat patch was firmly adhered to the skin and fastened by an elastic tubular net bandage (Elastofix, Insfarma, Germany). This process took approximately 1-min and this time was subtracted from the final race time of each participant.

Within 1-min of the end of the race, participants went to a finish area and body mass and body bioelectrical impedance were immediately measured using the same apparatus described previously. Participants were instructed to avoid drinking from the finish line till the post-race weighing and an experimenter assured compliance. Then, participants performed two countermovement vertical jumps and the whole-body isometric muscle strength test, as previously described. These performance tests were completed within 5-min of the end of the race. Participants then rested for 5-min and a venous blood sample was obtained. During this resting period, the sweat patches were removed using clean tweezers and placed in a sterile 10 mL- tube. Sweat patches that were detached from the skin or presented a leak were discarded.

After these protocols, the rate of perceived exertion during the race was self-rated using the Borg scale (6 to 20 points) while perceived leg muscle soreness was self-rated using a visual analog scale (0 to 10 points). Participants also filled out a detailed questionnaire about fluid and food intake during the race. Data on this questionnaire were used to calculate fluid, calorie and carbohydrate intake during the race. With this self-reported questionnaire, we also calculated electrolyte intake during the race (apart from the salt ingested with the capsule treatment). Finally, participants reported any incident during the intake of the capsules and the side-effects derived from their ingestion.

Blood and sweat sample analysis The blood was allowed to clot in situ and serum was separated by centrifugation (10 min at 5000 g) and frozen at -80ºC until the day of analysis. At a later date, the serum portion was analyzed for osmolality (1249, Advance 3MO, Spain), sodium, chloride, potassium and magnesium concentrations (Nova 16, NovaBiomedical, Spain). In addition, the serum creatine kinase concentration was measured as a blood marker of muscle damage by means of an autoanalyzer (AU5400, Beckman Coulter, US). The sweat was separated from the patches by centrifugation (10 min at 3000 g), transferred to 5-mL sealed tubes and refrigerated at 4 ºC. At a later date (within 2 days of the race), sweat osmolality was measured with the same osmometer employed for the serum samples while sweat electrolyte concentration were measured using an ion selective electrode analyzer (Cobas 6000, Roche, Madrid, Spain).

Statistical Analysis The normality of each variable was initially tested with the Shapiro-Wilk test. All the variables presented a normal distribution. For the variables obtained once during the experiment (race time, body mass change, sweat electrolyte concentration, self-rated fatigue and muscle soreness, etc) the comparison between groups (salt vs control) was performed using Student's t test for independent samples. For the variables obtained twice during the experiment (body mass, blood variables, jump performance, etc) the comparison between groups was performed by using a mixed model ANOVA (time × treatment) with repeated measures for the variable time. The data were analyzed with the statistical package SPSS version 19.0 (SPSS Inc., Chicago, IL). The significance level was set at P < 0.05. Data are presented as mean ± SD.

ELIGIBILITY:
Inclusion Criteria:

-Triathletes with previous experience in half-ironman

Exclusion Criteria:

-Potential participants (triathletes) with a previous history of muscle disorder, cardiac or kidney disease or those taking medicines or supplements during the two prior weeks were discarded.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-06; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Triathlon race time | The experiment will be carried out in 1 day. This variable will be obtained in this unique experimental day.
  Participants will compete in a real half-ironman triathlon and race time will be measured by means of chip timing. The chip timing will be adjusted in the participants's shoe.
  Race time will be measured in seconds.
Changes in blood parameters before and after the race | The experiment will be carried out in 1 day. This variable will be obtained in this unique experimental day
  The serum portion of each blood sample will be analyzed for osmolality (1249, Advance 3MO, Spain), sodium, chloride, potassium and magnesium concentrations (Nova 16, NovaBiomedical, Spain). ). In addition, the serum creatine kinase concentration will be measured as a blood marker of muscle damage by means of an autoanalyzer (AU5400, Beckman Coulter, US).
  Blood concentration (in mM) will be determined for each variable.
Sweat samples analysis | The experiment will be carried out in 1 day. This variable will be obtained in this unique experimental day
  The sweat will be obtained with sweat patches (Tegaderm 3m) and it will be separated from the patches by centrifugation (10 min at 3000 g), transferred to 5-mL sealed tubes and refrigerated at 4 ºC. At a later date (within 2 days of the race), sweat osmolality will be measured with the same osmometer employed for the serum samples while sweat electrolyte concentration were measured using an ion selective electrode analyzer (Cobas 6000, Roche, Madrid, Spain).
  Sweat electrolyte concentration will be measured in mM.

SECONDARY OUTCOMES:
Changes in total body water content (pre and post-race) | The experiment will be carried out in 1 day. This variable will be obtained in this unique experimental day
  Just 15-min before the race (and after their habitual warm-up), participants will be weighed in their competition clothes (without wetsuit) and a segmental bioelectrical impedance analysis will be performed (BC-418, Tanita, Japan) to predict pre-to-post race total body water changes.
  Total body water will be measured in kg.
Changes in whole body isometric force from pre to post-race | The experiment will be carried out in 1 day. This variable will be obtained in this unique experimental day
  Before and just after the race, whole-body isometric muscle strength will be measured by means of a hand-held pull gauge (Isocontrol Isométrico, EV-Pro, Spain) set at a frequency of 1000 Hz. For this measurement, participants will stand on a 50 × 50 cm iron base connected to a handle-bar by a non-elastic cable. The isometric gauge will be inserted within the cable and the height of the cable was individually set to provide a 135º knee flexion while the back and the arms will be completely extended. An adjustable lumbar-back protector was used for support and protection during the execution. Maximal and mean isometric strength were obtained during the test. Participants will be previously familiarized with this measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Del Coso, PhD, Principal Investigator — Camilo Jose Cela University
Locations (1):
- Exercise Physiology Laboratory, Camilo Jose Cela University, Villanueva de la Cañada, Madrid, Spain

REFERENCES:
- [Derived] Del Coso J, Gonzalez-Millan C, Salinero JJ, Abian-Vicen J, Areces F, Lledo M, Lara B, Gallo-Salazar C, Ruiz-Vicente D. Effects of oral salt supplementation on physical performance during a half-ironman: A randomized controlled trial. Scand J Med Sci Sports. 2016 Feb;26(2):156-64. doi: 10.1111/sms.12427. Epub 2015 Feb 14. PMID 25683094